CLINICAL TRIAL: NCT03155165
Title: Retroview™ vs. Conventional Colonoscopy: it is Time to Change?
Brief Title: Retroview™ Colonoscope and Lesion Detection Rate
Status: Completed | Type: Observational
Sponsor: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Responsible Party: Sponsor
Other Study IDs: DEC-19-2016
Record Dates: First submitted 2016-12-19; First posted 2017-05-16 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Colonic Neoplasms
Keywords: Colonoscopy, Retroview™ colonoscope, retrofex colonoscopy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Histology sample of polypectomies
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group A Retroview™ colonoscope: Patients that have a polyp already seen in a previous colonoscopy and the colonoscopy is indicated for polypectomy will be submitted to a Retroview™ colonoscope
  Interventions: Device: Retroview™ colonoscope
- Group B Retroview™ colonoscope: The rest of colonoscopies indicated will be submitted to a Retroview™ colonoscope
  Interventions: Device: Retroview™ colonoscope

INTERVENTIONS:
Device: Retroview™ colonoscope — The colonoscopy will be performed twice, with 2 different scopes, in tandem, by 2 endoscopists trained on retroflex withdrawal. First a conventional HD colonoscope with I-Scan will be used following the standard withdrawal technique and then the second endoscopist blinded to the first colonoscopy results, will perform the second colonoscopy using the Retroview™ scope with a combining withdrawal (retroflexed + standard withdrawal). The endoscopist that will perform each colonoscopy will be chosen randomly. After the examination, the endoscopist will fill a questionnaire detailing each polyp / adenoma found including the size and location.

SUMMARY:
Colonoscopy is considered the gold standard for colorectal polyp and cancer detection. However, even meticulous colonoscopy substantial numbers of colorectal polyps may be missed and carcinomas may not be prevented. Previous studies have found a 12-28% of miss rate for all polyps, a 31% for hyperplastic polyps and 6-27% for adenomas, with the higher miss rates noted for smaller polyps. The lesions missing rate depends on several factors as the location on difficult areas to be evaluated with conventional colonoscopes (the proximal side of the ileocecal valve, haustral folds, flexures or rectal valves), a flat shape, a poor bowel preparation and inadequate endoscopy technique, particularly rapid colonoscope withdrawal. Using the commonly available 140º angle of view colonoscope, approximately 13% of the colonic surface is unseen. The incorporation of colonoscopes with a 170-degree wide angled could not improve adenoma detection rate. The introduction of high definition (HD) colonoscopes and visual image enhancement technologies as narrow band imaging (NBI, Olympus America, Center Valley, PA), i-SCAN™ (PENTAX of America, Montvale, NJ) and Fuji Intelligent Chromo-Endoscopy (FICE™, Fujinon Endoscopy, Wayne, NJ) have improved the lesion characterization, but several studies proved no increase in adenoma detection rates. The Third Eye Retroscope (Avantis Medical Systems, Sunnyvale, CA) is a disposable retrograde viewing device advanced via the accessory channel of a standard colonoscope. Allows retrograde views behind colonic folds and flexures simultaneously with the forward view of the colon. Although it was shown an increase in adenoma detection rate by 11%-25%, it has many disadvantages. It requires a separate processor and the device is disposable making the cost bigger. Occupies the working channel of the colonoscope which limits the ability to suction. If a polyp is seen the viewing device has to be removed in order to perform the polypectomy. The optic is not high definition and finally, the endoscopist has to get used to visualizing and processing two simultaneous video streams from the colonoscope and from the retroscope device.

DETAILED DESCRIPTION:
The Retroview™ (PENTAX Medical, HOYA Co.) colonoscope has a short turning radius at the colonoscope tip, that allows a retroflexed view of the colon during withdrawal. This may allow for detection of polyps hidden behind flexures, folds and valves, from the cecum to the rectum. It offers many advantages like the ability to provide high definition views of the proximal aspects of colonic folds, flexures and valves with no additional equipment or device costs. The image is high definition and the colonoscope also incorporates i-SCAN technology. The suction/work channel of the colonoscope is available for therapeutic procedures. Polypectomy can be performed with the colonoscope in retroflexion, without losing views of the polyp. The only disadvantages are the higher consumed withdrawal time because the additional retroflexed withdrawal to the standard withdrawal and that a small portion of the colon is obscured by the shaft of the colonoscope in retroflexion that may be the reason why combined standard withdrawal with retroflexed withdrawal has proved to be better than retroflexed withdrawal alone.

The aim of this study is to determinate and compare the polyp / adenoma detection rate and lesion miss rate by performing a colonoscopy using conventional scopes vs PENTAX RetroView™ scope. As a secondary outcome, size of lesions will be measure in order to determinate if there is a difference between both technics.

MATERIALS AND METHODS

Setting: Instituto Ecuatoriano de Enfermedades Digestivas (IECED), Omni Hospital Academic Tertiary Center. We will include patients from December 2016 to July 2017. The study protocol and consent form has been approved by the Institutional Review Board and will be conducted according to the declaration of Helsinki. Patients will sign an informed consent.

Intervention: endoscopic technique The colonoscopy will be performed, in all cases, twice with 2 different scopes. One is a conventional HD colonoscope with I-Scan, tube diameter of 13.2 mm and total length 2023 mm (standard EC 3490LK, PENTAX, Montvale, NJ) and the other is the Retroview™ colonoscope with tube diameter of 11.6 mm and total length 2023 mm (EC-3490TLi, PENTAX, Montvale, NJ). The endoscopy images will be seen on a 27-inch, flat panel, HD LCD monitor (Radiance™ ultra SC-WU27-G1520 model). All of the participants will follow the same colonic preparation with 4 liters of polyethylene glycol (PEG) the day before and the bowel preparation will be evaluated using the Boston Bowel Preparation Scale. Two trained endoscopists on retroflex withdrawal will perform the colonoscopies. Both colonoscopies will be performed in tandem. First one endoscopist will perform the conventional colonoscopy using standard withdrawal technique and then the second endoscopist blinded to the first colonoscopy results, will perform the second colonoscopy with the Retroview scope and combination withdrawal (retroflexed + standard withdrawal). The endoscopist that will perform each colonoscopy will be chosen randomly. The minimum withdrawal time of 6 minutes that is recommended in literature will be respected in both cases. After the examination, the endoscopist will fill a questionnaire detailing each polyp / adenoma found including the size and location. The withdrawal time will be measured in both colonoscopies.

Statistical analysis: Baseline characteristics will be analyzed using Chi-square o Fisher Test for categorical variable and Mann-Whitney Test for continuing variables. If there are more than one polyp in one patients it will be considered individually for statistical purposes. A P value of less than 0.05 will be considered to be statistically significant. All the statistical analysis will be performed using SPSS software suite v.22.

Limitations: The protocol will be performed in only one center and by two endoscopists. There is no control group because the intention is to compare two endoscopy methods in the same setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients that agree to participate in the study.
* Able to understand and provide written informed consent.
* Colonoscopy indication for colorectal neoplasia screening or polyp surveillance.
* Colonoscopy indication for polypectomy.
* Colonoscopy indication for diagnostic workup including anemia, abdominal pain, constipation, abnormal imaging.

Exclusion Criteria:

* Age under 18 and over 80 years' old.
* Pregnancy
* Patients with heart disease, kidney, liver or severe metabolic disorder, who cannot tolerate sedation.
* Severe uncontrolled coagulopathy.
* Patients with difficulty understanding instructions of bowel preparation.
* Prior history of colon resection.
* Patients with an ileostomy or a colostomy.
* Abdomen or pelvis radiation therapy.
* Known inflammatory bowel disease, polyposis syndrome or acute diverticulitis.
* Suspected colonic obstruction or history of previous obstruction.
* Gastrointestinal bleeding.
* Lack of acceptance by the patient.
* Bowel preparation will be evaluated using the Boston Bowel Preparation Scale. Patients with < 2 points in at least one of the three segments of the colon (rectum plus left-side colon, transverse colon plus left and right flexure, right-side colon) will be excluded from statistical analysis as well as those who after the beginning of the colonoscopy, had to be aborted because of an inability to reach the cecum by unfavorable anatomy or impassable tumors / stenosis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the gastroenterology unit (IECED). All of the participants will have a clear colonoscopy indication. Group A will include patients that have a polyp already seen in a previous colonoscopy and the colonoscopy is indicated for polypectomy. Group B will include the rest of indicated colonoscopies. The distribution in groups A and B is with no intention to compeer the groups but in order to avoid a bias because the patients already have a known lesion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Polyp detection rate with the standard colonoscope and Retroview™ scope. | 8 month
  Polyps found with standard colonoscope / total of polys found X 100; polyps found with Retroview™ scope / total of polys found X 100; The total of polyps found will be determinated by the combination of both technics (standard colonoscope and Retroview™ scope)
Adenoma detection rate with the standard colonoscope and Retroview™ scope. | 8 month
  Adenomas found with standard colonoscope / total of adenomas found X 100; adenomas found with Retroview™ scope / total of adenomas found X 100. The total of adenomas found will be determinated by the combination of both technics (standard colonoscope and Retroview™ scope)

SECONDARY OUTCOMES:
Lesion miss rate with the standard colonoscope and Retroview™ scope. | 8 month
  Lesion miss rate: lesions missed / total of lesions (polyps and adenomas) X 100
Number and size of lesions (adenomas and polyps) detected with the standard colonoscope and Retroview ™ scope. | 8 month
  The number and size of lesions will be described in each patient with both procedures. The size will be measure using a standard biopsy catheter as comparison method.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Robles-medranda, MD, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Omnihospital, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Winawer SJ, Zauber AG, Ho MN, O'Brien MJ, Gottlieb LS, Sternberg SS, Waye JD, Schapiro M, Bond JH, Panish JF, et al. Prevention of colorectal cancer by colonoscopic polypectomy. The National Polyp Study Workgroup. N Engl J Med. 1993 Dec 30;329(27):1977-81. doi: 10.1056/NEJM199312303292701. PMID 8247072
- [Result] Hixson LJ, Fennerty MB, Sampliner RE, Garewal HS. Prospective blinded trial of the colonoscopic miss-rate of large colorectal polyps. Gastrointest Endosc. 1991 Mar-Apr;37(2):125-7. doi: 10.1016/s0016-5107(91)70668-8. PMID 2032595
- [Result] Heresbach D, Barrioz T, Lapalus MG, Coumaros D, Bauret P, Potier P, Sautereau D, Boustiere C, Grimaud JC, Barthelemy C, See J, Serraj I, D'Halluin PN, Branger B, Ponchon T. Miss rate for colorectal neoplastic polyps: a prospective multicenter study of back-to-back video colonoscopies. Endoscopy. 2008 Apr;40(4):284-90. doi: 10.1055/s-2007-995618. PMID 18389446
- [Result] Pickhardt PJ, Nugent PA, Mysliwiec PA, Choi JR, Schindler WR. Location of adenomas missed by optical colonoscopy. Ann Intern Med. 2004 Sep 7;141(5):352-9. doi: 10.7326/0003-4819-141-5-200409070-00009. PMID 15353426
- [Result] Robertson DJ, Greenberg ER, Beach M, Sandler RS, Ahnen D, Haile RW, Burke CA, Snover DC, Bresalier RS, McKeown-Eyssen G, Mandel JS, Bond JH, Van Stolk RU, Summers RW, Rothstein R, Church TR, Cole BF, Byers T, Mott L, Baron JA. Colorectal cancer in patients under close colonoscopic surveillance. Gastroenterology. 2005 Jul;129(1):34-41. doi: 10.1053/j.gastro.2005.05.012. PMID 16012932
- [Result] Bressler B, Paszat LF, Vinden C, Li C, He J, Rabeneck L. Colonoscopic miss rates for right-sided colon cancer: a population-based analysis. Gastroenterology. 2004 Aug;127(2):452-6. doi: 10.1053/j.gastro.2004.05.032. PMID 15300577
- [Result] Miller RE, Lehman G. Polypoid colonic lesions undetected by endoscopy. Radiology. 1978 Nov;129(2):295-7. doi: 10.1148/129.2.295. PMID 704840
- [Result] Soetikno RM, Kaltenbach T, Rouse RV, Park W, Maheshwari A, Sato T, Matsui S, Friedland S. Prevalence of nonpolypoid (flat and depressed) colorectal neoplasms in asymptomatic and symptomatic adults. JAMA. 2008 Mar 5;299(9):1027-35. doi: 10.1001/jama.299.9.1027. PMID 18319413
- [Result] Froehlich F, Wietlisbach V, Gonvers JJ, Burnand B, Vader JP. Impact of colonic cleansing on quality and diagnostic yield of colonoscopy: the European Panel of Appropriateness of Gastrointestinal Endoscopy European multicenter study. Gastrointest Endosc. 2005 Mar;61(3):378-84. doi: 10.1016/s0016-5107(04)02776-2. PMID 15758907
- [Result] East JE, Saunders BP, Burling D, Boone D, Halligan S, Taylor SA. Surface visualization at CT colonography simulated colonoscopy: effect of varying field of view and retrograde view. Am J Gastroenterol. 2007 Nov;102(11):2529-35. doi: 10.1111/j.1572-0241.2007.01429.x. Epub 2007 Jul 19. PMID 17640320
- [Result] Rex DK, Cutler CS, Lemmel GT, Rahmani EY, Clark DW, Helper DJ, Lehman GA, Mark DG. Colonoscopic miss rates of adenomas determined by back-to-back colonoscopies. Gastroenterology. 1997 Jan;112(1):24-8. doi: 10.1016/s0016-5085(97)70214-2. PMID 8978338
- [Result] McGill SK, Kothari S, Friedland S, Chen A, Park WG, Banerjee S. Short turn radius colonoscope in an anatomical model: retroflexed withdrawal and detection of hidden polyps. World J Gastroenterol. 2015 Jan 14;21(2):593-9. doi: 10.3748/wjg.v21.i2.593. PMID 25593483
- [Result] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102
- [Result] Rex DK, Petrini JL, Baron TH, Chak A, Cohen J, Deal SE, Hoffman B, Jacobson BC, Mergener K, Petersen BT, Safdi MA, Faigel DO, Pike IM. Quality indicators for colonoscopy. Gastrointest Endosc. 2006 Apr;63(4 Suppl):S16-28. doi: 10.1016/j.gie.2006.02.021. No abstract available. PMID 16564908
- [Result] Rex DK, Chadalawada V, Helper DJ. Wide angle colonoscopy with a prototype instrument: impact on miss rates and efficiency as determined by back-to-back colonoscopies. Am J Gastroenterol. 2003 Sep;98(9):2000-5. doi: 10.1111/j.1572-0241.2003.07662.x. PMID 14499778
- [Result] Fatima H, Rex DK, Rothstein R, Rahmani E, Nehme O, Dewitt J, Helper D, Toor A, Bensen S. Cecal insertion and withdrawal times with wide-angle versus standard colonoscopes: a randomized controlled trial. Clin Gastroenterol Hepatol. 2008 Jan;6(1):109-14. doi: 10.1016/j.cgh.2007.10.009. Epub 2007 Dec 11. PMID 18065277
- [Result] Deenadayalu VP, Chadalawada V, Rex DK. 170 degrees wide-angle colonoscope: effect on efficiency and miss rates. Am J Gastroenterol. 2004 Nov;99(11):2138-42. doi: 10.1111/j.1572-0241.2004.40430.x. PMID 15554993
- [Result] Chung SJ, Kim D, Song JH, Park MJ, Kim YS, Kim JS, Jung HC, Song IS. Efficacy of computed virtual chromoendoscopy on colorectal cancer screening: a prospective, randomized, back-to-back trial of Fuji Intelligent Color Enhancement versus conventional colonoscopy to compare adenoma miss rates. Gastrointest Endosc. 2010 Jul;72(1):136-42. doi: 10.1016/j.gie.2010.01.055. Epub 2010 May 20. PMID 20493487
- [Result] Nagorni A, Bjelakovic G, Petrovic B. Narrow band imaging versus conventional white light colonoscopy for the detection of colorectal polyps. Cochrane Database Syst Rev. 2012 Jan 18;1(1):CD008361. doi: 10.1002/14651858.CD008361.pub2. PMID 22258983
- [Result] Jin XF, Chai TH, Shi JW, Yang XC, Sun QY. Meta-analysis for evaluating the accuracy of endoscopy with narrow band imaging in detecting colorectal adenomas. J Gastroenterol Hepatol. 2012 May;27(5):882-7. doi: 10.1111/j.1440-1746.2011.06987.x. PMID 22098192
- [Result] Waye JD, Heigh RI, Fleischer DE, Leighton JA, Gurudu S, Aldrich LB, Li J, Ramrakhiani S, Edmundowicz SA, Early DS, Jonnalagadda S, Bresalier RS, Kessler WR, Rex DK. A retrograde-viewing device improves detection of adenomas in the colon: a prospective efficacy evaluation (with videos). Gastrointest Endosc. 2010 Mar;71(3):551-6. doi: 10.1016/j.gie.2009.09.043. Epub 2009 Dec 16. PMID 20018280
- [Result] Leufkens AM, DeMarco DC, Rastogi A, Akerman PA, Azzouzi K, Rothstein RI, Vleggaar FP, Repici A, Rando G, Okolo PI, Dewit O, Ignjatovic A, Odstrcil E, East J, Deprez PH, Saunders BP, Kalloo AN, Creel B, Singh V, Lennon AM, Siersema PD; Third Eye Retroscope Randomized Clinical Evaluation [TERRACE] Study Group. Effect of a retrograde-viewing device on adenoma detection rate during colonoscopy: the TERRACE study. Gastrointest Endosc. 2011 Mar;73(3):480-9. doi: 10.1016/j.gie.2010.09.004. Epub 2010 Nov 10. PMID 21067735
- [Result] Hewett DG, Rex DK. Miss rate of right-sided colon examination during colonoscopy defined by retroflexion: an observational study. Gastrointest Endosc. 2011 Aug;74(2):246-52. doi: 10.1016/j.gie.2011.04.005. Epub 2011 Jun 15. PMID 21679946